CLINICAL TRIAL: NCT06644898
Title: The Effect of Aerobic Exercise Training at Different Slope Types on Balance in COPD Patients
Brief Title: The Effect of Gait Training Using Different Slope Types on Balance in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Meryem BEKTAŞ KARAKUŞ, Research Assistant, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-11/491
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: aerobic exercise, slope, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level walking (Active Comparator): It will walk at a 0-degree slope (0) throughout the research.
  Interventions: Other: Level walking training
- Downhill walking (Experimental): It will walk at a 10-degree downhill slope (-10) throughout the research.
  Interventions: Other: Downhill walking training
- Uphill walking (Experimental): It will walk at a 10-degree uphill slope (+10) throughout the research.
  Interventions: Other: Uphill walking training

INTERVENTIONS:
Other: Level walking training — For 8 weeks, level walking training will be done 2 times a week at a slope of 0 degrees.
  Arms: Level walking
Other: Downhill walking training — For 8 weeks, downhill walking training will be done 2 times a week at a slope of -10 degrees.
  Arms: Downhill walking
Other: Uphill walking training — For 8 weeks, uphill walking training will be done 2 times a week at a slope of +10 degrees.
  Arms: Uphill walking

SUMMARY:
Although COPD is basically a respiratory system disease, its effects are not limited to the respiratory system. In this context, one parameter affected in COPD patients is balance. Recent studies have highlighted the importance of assessing balance and incorporating it into treatment options such as pulmonary rehabilitation. In this context, we aim to diversify the training by using different slope types (downhill, level, uphill) in aerobic exercise training, which is a strong component of pulmonary rehabilitation, and to evaluate the effect of slope type on balance. Testing different types of inclines in aerobic exercise training has the potential to result in different muscular gains. We anticipate that this may result in different balance gains.

DETAILED DESCRIPTION:
The convenience sampling method will be used as the sampling method in the research.

In this study, sample size was calculated by a priori power analysis using G*Power 3.1.9.4 software. In the analysis for analysis of variance (ANOVA: repeated measures, between factors) with two factors and repeated measures; effect size f = 0.62 (based on data obtained from previous study, Borghi-Silva et al, 2009), significance level α = 0.05, statistical power (1 - β) = 0.80, number of groups 3, number of measures 2 and correlation coefficient between measures r = 0.5. According to the calculation, it was predicted that the study would reach sufficient statistical power with a total of 24 participants, 8 participants in each group.

There will be three groups in the study: downhill walking, uphill walking, and level walking. The downhill walking and uphill walking groups will be included as the study group and the level walking group will be included as the control group. Participants will be distributed equally to the three groups. Patients will be assigned to these groups by block randomization method using https://www.randomizer.org/ website.

All three groups will be administered a 6-minute walking test at baseline, and participants will be subjected to a common 8-week, twice-weekly treadmill walking training program in which the speed is determined and increased according to the average speed they walk in this test, and in addition to this, the duration is also increased. One session of the training program will consist of warming up, loading, and cooling down on the treadmill.

During the training, the slope of the treadmill will be adjusted to +10 degrees for uphill walking, -10 degrees for downhill walking, and 0 degrees for level walking and will be kept constant for 8 weeks. A special wooden wedge apparatus will be made under the normal treadmill to give -10 downhill slope.

Primary outcome measurements will be made at baseline and at the end of week 8.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD (A, B, E groups according to GOLD assessment)
* Ambulate on your own
* Not having any contraindications for exercise

Exclusion Criteria:

* Being in GOLD 4 stage in spirometric evaluation
* Presence of hypoxemia
* Participation in another pulmonary rehabilitation program within the last 6 months
* Having an exacerbation in the last 1 month
* Being diagnosed with additional respiratory disease (asthma, bronchiectasis, etc.)
* Having had pulmonary surgery
* Having an orthopedic, neurological or cardiac disease that affects exercise
* Having uncontrolled hypertension or diabetes
* Presence of malignancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postural stability test | Up to 8 weeks.
  The test reflects a person's ability to maintain the center of balance.
Limits of Stability (LOS) Test | Up to 8 weeks.
  The maximum vertical angle that the body can reach while standing without losing balance is called the stability limit.
Clinical Test of Sensory Integration of Balance (CTSIB) | Up to 8 weeks.
  The test assesses how well the person can integrate sensory input to maintain balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Department of Physiotherapy and Rehabilitation, Istanbul, Eyüp Sultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Borghi-Silva A, Arena R, Castello V, Simoes RP, Martins LE, Catai AM, Costa D. Aerobic exercise training improves autonomic nervous control in patients with COPD. Respir Med. 2009 Oct;103(10):1503-10. doi: 10.1016/j.rmed.2009.04.015. Epub 2009 May 22. PMID 19464865
- [Background] Loughran KJ, Atkinson G, Beauchamp MK, Dixon J, Martin D, Rahim S, Harrison SL. Balance impairment in individuals with COPD: a systematic review with meta-analysis. Thorax. 2020 Jul;75(7):539-546. doi: 10.1136/thoraxjnl-2019-213608. Epub 2020 May 14. PMID 32409612
- [Background] Kaygusuz MH, Oral Tapan O, Tapan U, Genc S. Balance impairment and cognitive dysfunction in patients with chronic obstructive pulmonary disease under 65 years. Clin Respir J. 2022 Mar;16(3):200-207. doi: 10.1111/crj.13469. Epub 2022 Jan 26. PMID 35081270
- [Background] Jirange P, Vaishali K, Sinha MK, Bairapareddy KC, Alaparthi GK. A Cross-Sectional Study on Balance Deficits and Gait Deviations in COPD Patients. Can Respir J. 2021 Jan 6;2021:6675088. doi: 10.1155/2021/6675088. eCollection 2021. PMID 33505539
- [Background] Eymir M, Yakut H, Ozalevli S, Alpaydin AO. Static and dynamic balance impairment and relationship with disease-related factors in patients with chronic obstructive pulmonary disease : A cross-sectional study. Wien Klin Wochenschr. 2021 Nov;133(21-22):1186-1194. doi: 10.1007/s00508-021-01918-8. Epub 2021 Aug 5. PMID 34351502
- [Background] Alexander N, Strutzenberger G, Ameshofer LM, Schwameder H. Lower limb joint work and joint work contribution during downhill and uphill walking at different inclinations. J Biomech. 2017 Aug 16;61:75-80. doi: 10.1016/j.jbiomech.2017.07.001. Epub 2017 Jul 11. PMID 28734544